CLINICAL TRIAL: NCT07219511
Title: A Safety, Tolerability, and Biomarker Trial of VS-041 in Participants With Heart Failure With Preserved Ejection Fraction (HFpEF)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vasa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VS-041-102
Record Dates: First submitted 2025-10-17; First posted 2025-10-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Heart; Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Heart Failure with Preserved Ejection Fraction; HFpEF

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Low Dose VS-041 (Experimental)
  Interventions: Drug: VS-041
- High Dose VS-041 (Experimental)
  Interventions: Drug: VS-041

INTERVENTIONS:
Drug: VS-041 — VS-041 high dose, VS-041 low dose or Placebo tablet BID
  Arms: High Dose VS-041; Low Dose VS-041
Other: Placebo — Placebo to match VS-041
  Arms: Placebo

SUMMARY:
A Safety, Tolerability, and Biomarker Trial of VS-041 in Participants with Heart Failure with Preserved Ejection Fraction (HFpEF)

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all inclusion criteria to be eligible for trial participation.

1. Males or females ≥ 50 years of age at the time of signing the informed consent.
2. Diagnosis of HFpEF as defined by European Society of Cardiology or American College of Cardiology/American Heart Association criteria
3. NYHA Functional Class II or III
4. LVEF ≥ 50% demonstrated by echocardiography (ECHO) performed at Screening and evidence of heart failure with history of at least one HF hospitalization
5. Elevated NT-proBNP at Screening
6. NordicPRO-C6™ ≥ 11 ng/mL at Screening.
7. Stable dose of all concomitant HF medications for at least 4 weeks prior to Screening.
8. Body weight of at least 110 lbs (50 kg) and body mass index (BMI) within the range ≥ 18 to < 45 kg/m2.
9. Males must agree to the contraception requirements and females must be of non-childbearing potential
10. Able to understand and willing to sign a written informed consent form (ICF).
11. Willing and able to comply with trial procedures and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Female trial participant who is pregnant or breastfeeding.
2. Known hypersensitivity to VS-041.
3. Cardiovascular disease other than HFpEF
4. Active intercurrent illness such as acute bacterial or viral infection.
5. History of illicit drug or alcohol abuse or addiction that in the opinion of the PI could affect participation.
6. Serologic evidence of Hepatitis B or Hepatitis C or human immunodeficiency virus (HIV) at Screening.
7. Acute decompensated HF within 30 days of Screening
8. Lung disease within 12 months prior to Screening
9. History of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years.
10. History of any other condition including psychiatric disorders that, in the opinion of the PI, may preclude the participant from following and completing the protocol.
11. Have participated within the last 6 months in a clinical study involving an investigational product.
12. Any other reason which, in the opinion of the PI, would prevent the participant from participating in the trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Participant incidence of treatment-emergent adverse events (TEAEs) | From Baseline to Day 28
  To evaluate the safety and tolerability of VS-041 in participants with HFpEF
Change from baseline over time in serum NordicPRO-C6 | From Baseline to Day 28
  To evaluate the impact of VS-041 on key biomarkers in participants with HFpEF
Change from baseline over time in serum endotrophin | From Baseline to Day 28
  To evaluate the impact of VS-041 on key biomarkers in participants with HFpEF
Change from baseline over time in serum NT-proBNP | From Baseline to Day 28
  To evaluate the impact of VS-041 on key biomarkers in participants with HFpEF

SECONDARY OUTCOMES:
Pharmacokinetic profiles and parameters derived for VS-041 - Tmax | From Baseline to Day 28
  To assess PK of twice-daily VS-041 in participants with HFpEF
Pharmacokinetic profiles and parameters derived for VS-041 - Cmax | From Baseline to Day 28
  To assess PK of twice-daily VS-041 in participants with HFpEF

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - National Institute of Clinical Research, Huntington Beach, California
  - FOMAT, Santa Maria, California
  - Invivocure LLC, Van Nuys, California
  - New Generation of Medical Research, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Amavita Health, North Miami Beach, Florida
  - Chicago Medical Research, Hazel Crest, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Louisiana Heart Center, Slidell, Louisiana
  - Washington University, St Louis, Missouri
  - Ash Research Clinic, Brick, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Wake Forest, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided